CLINICAL TRIAL: NCT05544383
Title: Effectiveness of an Interdisciplinary Pain Education Program in Public Health: a Pragmatic Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal University of Espirito Santo (Other)
Responsible Party: Principal Investigator, Valéria Valim, Professor, Federal University of Espirito Santo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUEspiritoSanto
Record Dates: First submitted 2022-09-14; First posted 2022-09-16 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Musculoskeletal Pain
Keywords: Health Education; Self Efficacy; Health-Related Quality Of Life; Functional Health Literacy
MeSH Terms: conditions — Musculoskeletal Pain; Health Education

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Interdisciplinary Pain Education Program and conventional physical therapy treatment
  Interventions: Behavioral: Interdisciplinary Pain Education Program; Other: Conventional Physiotherapy treatment
- Comparison group (Active Comparator): Conventional physical therapy treatment
  Interventions: Other: Conventional Physiotherapy treatment

INTERVENTIONS:
Behavioral: Interdisciplinary Pain Education Program — It is an operative group model, with the objective of promoting education in pain, where the patient occupies an active and central space in the learning process, with work focused on the dysfunctional beliefs of chronic pain, performing programmed tasks to promote autonomy in activities daily life and behavior change. The group works with one meeting per week, during the routine opening hours of the clinic, with each day a theme of a professional area being addressed, totaling 5 meetings, lasting approximately two hours.
  Arms: Intervention group
Other: Conventional Physiotherapy treatment — The therapeutic approach consists of rehabilitation methods and techniques, with the aim of restoring, developing and conserving the patient's physical capacity and functionality, including manual therapy and kinesiotherapy, in addition to the use of resources such as electrotherapy, thermotherapy and auriculotherapy. The treatment is performed at the Physiotherapy outpatient clinic, twice a week, with an average duration of 45 minutes, for a period that lasts an average of 10 sessions in clinical cases of chronic musculoskeletal pain.

SUMMARY:
The objective of this study is to evaluate the effectiveness of an interdisciplinary pain education program in improving self-efficacy and promoting quality of life in patients with chronic musculoskeletal pain in public health. This is a pragmatic clinical trial carried out with patients referred to the Physical Therapy sector of a municipality who will be allocated in an interdisciplinary pain education intervention group or a comparison group of conventional physical therapy treatment.

DETAILED DESCRIPTION:
his is a pragmatic clinical trial carried out with patients referred to the Physical Therapy sector of a municipality who will be allocated in an interdisciplinary pain education intervention group or a comparison group of conventional physical therapy treatment. Clinical characteristics of pain will be evaluated by multidimensional questionnaires, in addition to self-efficacy, quality of life, functional literacy and sociodemographic profile. Health professionals will be evaluated by an attitude towards pain inventory. It is expected to demonstrate the effectiveness of interdisciplinary pain education work in managing the biopsychosocial impacts of pain by promoting knowledge and self-management strategies in the care of this chronic condition. As it is a light and collective technology, it can reduce the burden of the disease and support public policy decision-making in the management of chronic pain in public health.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical picture of chronic musculoskeletal pain, aged over 18 years, being SUS users referred for Physiotherapy treatment.

Exclusion Criteria:

* Patients with a clinical picture of acute pain, post-traumatic or post-surgical pain, cancer pain and neuropathic pain, as well as those with autoimmune diseases. Patients with cognitive problems who cannot understand and respond to the questionnaires and who also have other physical disabilities unrelated to the chronic pain condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Pain Self-Efficacy Questionnaire | 2 weeks
  The total score is calculated by adding the scores for each of the 10 items, resulting in a value ranging from 0 to 60, with higher scores reflecting stronger self-efficacy beliefs.
Pain Self-Efficacy Questionnaire | 3 months
  The total score is calculated by adding the scores for each of the 10 items, resulting in a value ranging from 0 to 60, with higher scores reflecting stronger self-efficacy beliefs.

SECONDARY OUTCOMES:
Brief Pain Inventory | 2 weeks
  pain-related scores ranging from zero (did not interfere) to ten (completely interfered)
Brief Pain Inventory | 3 months
  pain-related scores ranging from zero (did not interfere) to ten (completely interfered)
EuroQol (EQ-5D-3L) | 2 weeks
  patient's quality of life through self-assessment in five dimensions: mobility; self-care; usual activities; pain/discomfort; anxiety / depression. Each dimension has 3 levels: no problems, some problems, extreme problems/disability
EuroQol (EQ-5D-3L) | 3 months
  patient's quality of life through self-assessment in five dimensions: mobility; self-care; usual activities; pain/discomfort; anxiety / depression. Each dimension has 3 levels: no problems, some problems, extreme problems/disability
Health Literacy Scale (HLS-14) | 2 weeks
  assesses the level of health literacy through fourteen questions on a five-point Likert scale, in three dimensions of literacy: functional and communicative with 5 items each, and critical with 4 items.
Health Literacy Scale (HLS-14) | 3 months
  assesses the level of health literacy through fourteen questions on a five-point Likert scale, in three dimensions of literacy: functional and communicative with 5 items each, and critical with 4 items.
Survey of Pain Attitudes-Professionals (IAD-Profissionais) | 1 day
  20 items, covering 6 domains: emotion, control, disability, solicitude, medical cure and physical harm

CONTACTS AND LOCATIONS:
Overall Officials: Valéria Valim, PhD, Principal Investigator — Federal University of Espirito Santo

IPD SHARING:
Plan to Share IPD: No